CLINICAL TRIAL: NCT06282640
Title: Comparıson Of Electromyography Results Before And After Vıtamın D Treatment In Patıents Wıth Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Ayşe Güç (Other Government)
Collaborators: Kayseri City Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Ayşe Güç, medical doctor, Kayseri Education and Research Hospital
Organization: Kayseri Education and Research Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 567
Record Dates: First submitted 2024-01-29; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Carpal Tunnel Syndrome; Vitamin D Deficiency
Keywords: Carpal Tunnel Syndrome; Vitamin D Deficiency; Electrophysiologia
MeSH Terms: conditions — Carpal Tunnel Syndrome; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D in Carpal Tunnel Syndrome (Experimental)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D replacement therapy was administered at 50,000 IU weekly for 8 weeks.

SUMMARY:
Therefore, we aimed to evaluate the effectiveness of vitamin D replacement therapy on pain, electrophysiological parameters, ultrasonographic measurement results and functional status scales in CTS patients with low serum vitamin D levels.

DETAILED DESCRIPTION:
Introduction: Apart from its effect on bone health, vitamin D is also known to have beneficial effects on the neurological system. In studies, vitamin D levels were found to be low in patients with Carpal Tunnel Syndrome (CTS). However, studies examining the effects of vitamin D replacement on CTS are limited. Therefore, we aimed to evaluate the effectiveness of vitamin D replacement therapy on pain, electrophysiological parameters, ultrasonographic measurement results and functional status scales in CTS patients with low serum vitamin D levels. Materials and Methods: Our study was planned as an observational and analytical prospective. Vitamin D loading therapy was given to patients with serum vitamin D levels below 20ng/ml and mild-moderate CTS detected by electroneuromyography (ENMG). Patients with vitamin D levels above 20 ng/ml after 8 weeks were included in the study. Each patient was given a rest splint and exercise program. Patients were evaluated before and 3 months after treatment with electrophysiological, ultrasonographic, VAS, pinch-grip strength, two-point discrimination, monofilament test and Boston symptom severity scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old male or female gender
* Those with mild to moderate CTS according to ENMG,
* Vitamin D level <20.

Exclusion Criteria:

* Severe CTS according to ENMG
* Thenar region atrophy
* diabetes mellitus,
* rheumatoid arthritis,
* hyperthyroidism,
* hypothyroidism
* Traumatic nerve injury, history of surgery
* Polyneuropathy
* Pregnancy
* Severe psychiatric illness
* Poor orientation and cooperation,
* Injection (corticosteroid, ozone, stem cell…) applied for CTS treatment within 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
electrophysiological scale. | at the baseline and immediately after treatment
  Electrophysiological Evaluation: Neurowerk (SIGMA-Medizin-TechnicGmbH/Germany) brand ENMG device was used. Patients were evaluated at room temperature of approximately 25 °C. All measurements were made by the same doctor. Our clinic's reference values for the diagnosis of CTS are shown below

SECONDARY OUTCOMES:
monofilament test | at the baseline and immediately after treatment
  Semmes-Weinstein monofilament test (SWMT): The first three fingertips on the palmar surface of the hand included with the 6-monofilament set of Baseline company were evaluated. Monofilament number 2.83 was taken as the threshold value for normal sensory value. SWMT was applied blindly by the same occupational therapist who was unaware of the patients' disease and the treatment they received.

OTHER OUTCOMES:
Boston symptom severity scale | at the baseline and immediately after treatment
  Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ): The questionnaire consists of two parts. "Boston Symptom Severity Scale (BSSS)", which questions the severity of symptoms, consists of 11 questions. "Boston Functional Status Scale (BFSS)", which evaluates functional capacity, consists of 8 questions. The degree of difficulty of symptoms and functional activity increases towards 5 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)